CLINICAL TRIAL: NCT07202546
Title: A Phase 2b Randomized, Open-Label Active Controlled Study Evaluating the Safety and Efficacy of Oral VH4524184 Coadministered With Emtricitabine and Tenofovir Alafenamide in Treatment Naive Viremic Persons With HIV-1 (INNOVATE Study)
Brief Title: A Phase 2b Study Evaluating Oral VH4524184 Regimens in Treatment Naïve Persons With HIV-1 (INNOVATE Study)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 222638; 2025-521918-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-30; First posted 2025-10-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: Fixed dose combination; Antiretroviral; Antiviral; Naive viremics; Innovate; VH4524184
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Racivir; tenofovir alafenamide; Tablets; emtricitabine tenofovir alafenamide; dolutegravir; Lamivudine

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VH4524184 Dose A+ FTC / TAF (Experimental): Participants receive a daily oral dose of VH4524184 Dose A (Low dose) in combination with a fixed dose containing FTC/TAF starting Day 1 until Month 12.
  Interventions: Drug: VH4524184; Drug: Emtricitabine (FTC) and tenofovir alafenamide (TAF) Fixed Dose Combination (FDC) tablets
- VH4524184 Dose B + FTC / TAF (Experimental): Participants receive a daily oral dose of VH4524184 Dose B (High dose) in combination with a fixed dose containing FTC / TAF beginning on Day 1 until the Month 12.
  Interventions: Drug: VH4524184; Drug: Emtricitabine (FTC) and tenofovir alafenamide (TAF) Fixed Dose Combination (FDC) tablets
- DTG + 3TC (Active Comparator): Participants receive a daily oral dose of DTG and 3TC (fixed dose combination) from Day 1 through Month 24.
  Interventions: Drug: Dolutegravir / Lamivudine (DTG/3TC)
- VH4524184 selected dose + FTC / TAF (Experimental): Participants receive a selected dose of VH4524184, combined with FTC/TAF, orally once daily from to Month 12 to Month 24.
  Interventions: Drug: VH4524184; Drug: Emtricitabine (FTC) and tenofovir alafenamide (TAF) Fixed Dose Combination (FDC) tablets

INTERVENTIONS:
Drug: VH4524184 — Oral tablet will be administered.
  Arms: VH4524184 Dose A+ FTC / TAF; VH4524184 Dose B + FTC / TAF; VH4524184 selected dose + FTC / TAF
Drug: Emtricitabine (FTC) and tenofovir alafenamide (TAF) Fixed Dose Combination (FDC) tablets — Oral table will be administered.
  Other Names: DESCOVY
  Arms: VH4524184 Dose A+ FTC / TAF; VH4524184 Dose B + FTC / TAF; VH4524184 selected dose + FTC / TAF
Drug: Dolutegravir / Lamivudine (DTG/3TC) — Oral tablets will be administered.
  Other Names: DOVATO
  Arms: DTG + 3TC

SUMMARY:
This clinical study is testing a new medication, VH4524184, to see if it can effectively treat HIV-1 in adults who have never received treatment for their infection. The study is comparing two different doses of VH4524184, each taken with the medications emtricitabine and tenofovir alafenamide (FTC/TAF), to a standard HIV treatment called dolutegravir and lamivudine (DTG/3TC). The purpose of the study is to provide data on the long-term antiviral activity of the VH4524184 and provide information regarding dosing formulation for further evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years of age (or older, if required for adults by local regulations) at the time of signing the informed consent.
2. Screening CD4+ T-cell count >200 cells/microlitre (µL).
3. Documented HIV-1 infection and Screening plasma HIV-1 RNA of ≥1000 copies/millilitre (mL). A single repeat of this test is allowed within a single Screening period to determine eligibility.
4. Treatment-naive: Defined as no ARVs (in combination or monotherapy) received after the diagnosis of HIV-1 infection.
5. Body weight >=50.0 kilogram (kg) [(110 pounds (lbs)] for participants assigned male at birth and >=45.0 kg (99 lbs) for participants assigned female at birth. BMI within the range 18.5-35.5 kg/m^2 (inclusive - applies to males and females).
6. There are no contraceptive requirements for participants assigned male at birth.
7. Participants assigned female at birth are eligible to participate if they are not pregnant or breastfeeding and one of the following conditions applies:

   * Is a Participant of non-childbearing potential (PONCBP);OR Is a Participant of childbearing potential (POCBP) and using a contraceptive method with a failure rate of less than (<) 1% prior to and during the study intervention period, and for at least 1 week after the last dose of VH4524184 plus FTC/TAF FDC, or through the end of study (if in the control arm and never received VH4524184).
   * A POCBP must have a negative pregnancy test at Screening (serum) and on Day 1 (urine) before the first dose of study intervention.
   * If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. Participant with a positive serum test must be excluded.
8. Capable of giving signed informed consent.

Exclusion Criteria:

1. Participants who are breastfeeding or plan to breastfeed during the study.
2. Participants with acute HIV infection, evidenced by acute retroviral syndrome (e.g., fever, malaise, fatigue, etc.) and/or evidence of recent (within 3 months) documented viremia without antibody production and/or evidence of recent (within 3 months) documented seroconversion.
3. Any evidence of an active Centres for Disease Control and Prevention (CDC) Stage 3 disease [CDC 2014], except cutaneous Kaposi's sarcoma not requiring systemic therapy during the study. Historical CD4+ cell counts less than 200 cells/µL are not exclusionary.
4. Unstable liver disease known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
5. History of cirrhosis with or without viral hepatitis co-infection.
6. Participants with HCV co-infection will be excluded from the study.
7. Individuals who are co-infected with HIV and HBV will be excluded Participants diagnosed with syphilis at Screening (i.e., positive syphilis testing) should be treated as per local guidelines and will be eligible to enroll at any time regardless of the stage of disease.
8. Uncontrolled malignancy is excluded, whereas participants who have controlled malignancies may be included in agreement between the investigator and the ViiV Healthcare medical monitor.
9. Any pre-existing physical, or mental condition (including alcohol or drug abuse) which, in the opinion of the investigator (with or without psychiatric evaluation) or the ViiV Healthcare medical monitor, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
10. Any condition which, in the opinion of the investigator or the ViiV Healthcare medical monitor, that may interfere with the absorption, distribution, metabolism or excretion of the study interventions or render the participant unable to take oral medication and normal gastrointestinal anatomy or motility or hepatic and/or renal function
11. Clinically significant CV disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
12. Participants receiving any protocol-prohibited medication and who are unwilling or unable to switch to an alternate medication.
13. History of sensitivity to any of the study medications, or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the investigator or ViiV Healthcare medical monitor, contraindicates their participation.
14. Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (≤325 mg) or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease.
15. Treatment with any of the following agents within 60 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, any systemic immune suppressant.
16. Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 30 days of Day 1.
17. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
18. Exposure to an approved vaccine within 14 days prior to Day 1.
19. Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research
20. Participants with known or suspected presence of virologic resistance mutations as defined by the Stanford HIV Drug Resistance Database to INSTIs or NRTIs. This determination will be based on local virologic resistance testing, either at Screening or within the 3 months prior to Screening. ViiV Healthcare clinical virologist and/or ViiV Healthcare medical monitor will verify eligibility to this criterion prior to Day 1.
21. Creatinine clearance (eGFR) of <60 mL/min/1.73 m2 via CKD-EPI race neutral method [Delgado, 2021].
22. ALT >3 times the upper limit of normal (ULN). A single repeat of ALT is allowed within a single screening period to determine eligibility.
23. Any Grade 4 laboratory abnormality at screening, except for a Grade 4 CPK and lipid abnormalities (e.g., total cholesterol, triglycerides, etc.) will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the ViiV Healthcare medical monitor. A single repeat of any lab abnormality is allowed within a single screening period to determine eligibility.
24. Any acute laboratory abnormality at screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
25. Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination and will be the screening ECG entered into the eCRF): QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 msec (males) or >470 msec (females); >480 msec for participants with bundle branch block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) Suppression (<50 copies/millilitre) as per FDA Snapshot Methodology | At Month 12

SECONDARY OUTCOMES:
Percentage of Participants Maintaining Plasma HIV-1 RNA Suppression (<50 copies/mL) Based on Observed Laboratory Results | Day 1 to Month 24
Percentage of Participants Achieving Plasma HIV-1 RNA Suppression (<50 copies/ml) as per FDA Snapshot Methodology | Day 1 to Month 24
Change From Baseline in Cluster of Differentiation 4 (CD4+) T-cell Counts | Day 1 to Month 24
  Blood samples will be collected for assessment of T-cells subsets (CD4+ T-cells count) by flow cytometry.
Number of Participants with Any Adverse Event (AE) | Day 1 to Month 24
Number of Participants with AEs by Severity | Day 1 to Month 24
  The severity will be assessed using The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) Version 2.1 where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening and Grade 5 = Death.
Number of Participants with AEs Leading to Study Treatment Discontinuation | Day 1 to Month 24
Plasma Concentration of VH4524184 | Day 1 to Month 24
  Blood samples will be collected at indicated time point for PK analysis of VH4524184.

IPD SHARING:
Plan to Share IPD: Yes
Sudy Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf